CLINICAL TRIAL: NCT02160717
Title: Beta-Cell Function in Young Turner Syndrome Patients
Brief Title: Risk of Diabetes in Young Turner Syndrome Patients
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCHMC-906; UL1TR000077 (NIH)
Record Dates: First submitted 2014-06-04; First posted 2014-06-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome; Diabetes
MeSH Terms: conditions — Turner Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Turner Syndrome: Female with Turner Syndrome
- Healthy Controls: Healthy Female

SUMMARY:
Turner Syndrome is a common genetic disorder. Seventy percent of adults with Turner Syndrome have abnormalities in glucose metabolism which can lead to diabetes. The current screening guidelines for diabetes in Turner Syndrome are not specific and involve a fasting blood sugar once a year. The objective of this study is to determine if there are abnormalities in glucose metabolism and pancreatic function in young girls with Turner Syndrome. The study hypothesis is that pancreatic dysfunction (specifically of the beta cells that make insulin) is more prevalent in girls with Turner Syndrome compared to healthy controls.

DETAILED DESCRIPTION:
The study will be conducted at Children's Hospital Medical Center, Cincinnati. The study will require 1 visit to the hospital where the subject will have an oral glucose tolerance test and a physical exam

ELIGIBILITY:
Turner Syndrome Females:

Inclusion Criteria:

* Turner Syndrome confirmed by chromosomal testing
* On standard therapy (growth hormone and or estrogen)

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* Polycystic Ovarian Syndrome
* Pregnancy
* On any medications that alter blood sugar

Healthy Female Controls:

Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* Polycystic Ovarian Syndrome
* Pregnancy
* On any medications that alter blood sugar

Ages: 6 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary Care Clinic Turner Syndrome Center of Cincinnati Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Beta-Cell Function measured as Disposition Index | 1 day at screening
  Disposition index will be calculated based on the results of the oral glucose tolerance test using minimal modeling (computer program)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Sheanon, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center, Cincinnati, Cincinnati, Ohio, United States